CLINICAL TRIAL: NCT04096105
Title: A Phase 1, Randomized, Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of CC-93538 in Healthy Japanese and Caucasian Adult Subjects
Brief Title: Japanese Pharmacokinetic Bridging Study for CC-93538
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CC-93538-CP-001; U1111-1238-7252 (Other: WHO)
Record Dates: First submitted 2019-09-04; First posted 2019-09-19 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy subjects; CC-93538; Japanese PK bridging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CC-93538 in Japanese subjects (Experimental): Twenty-four Japanese subjects will be randomized into 1 of 2 dose levels in a 1:1 fashion so that 12 subjects will receive a 180 mg or 360 mg dose via SC injection.
  Interventions: Drug: CC-93538
- Administration of CC-93538 in Caucasian subjects (Experimental): Twenty-four Caucasian subjects will be matched to Japanese subjects by weight (± 20%) and receive a 180 mg or 360 mg dose via SC injection
  Interventions: Drug: CC-93538

INTERVENTIONS:
Drug: CC-93538 — a single dose CC-93538 SC

SUMMARY:
This is an open-label, randomized, parallel design study to evaluate the PK, safety, tolerability and immunogenicity of single SC doses of CC-93538 in healthy Japanese and Caucasian adult subjects.

A total of approximately 48 subjects, 24 Japanese and 24 Caucasians, will be enrolled. Japanese subjects will be enrolled first and randomized 1:1 to receive a single SC dose of either 180 mg or 360 mg CC-93538. Caucasian subjects will then be enrolled and matched to Japanese subjects (1:1) by weight (± 20%) and receive the same single SC dose of either 180 mg or 360 mg CC-93538.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject must be male or non-pregnant female, aged ≥ 18 and ≤ 55 years of age at the time of signing the ICF.
2. Subject must have a body weight of at least 40 kg; a BMI ≥18 and ≤ 30 kg/m2 at screening. Japanese and Caucasian subjects will be matched by body weight (± 20%).
3. Japanese subjects must have been born in Japan and not have lived outside of Japan > 5 years, have both parents and grandparents of Japanese origin, and have not significantly modified their diets since leaving Japan.
4. Caucasian subjects must be of European or Latin American descent (ie, White).
5. Subject must be in good health, as determined by the Investigator on the basis of medical history, clinical laboratory safety test results, vital signs, 12-lead ECG, and PE at screening.
6. Female subjects not of childbearing potential must:

   1. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before Screening, or
   2. Postmenopausal (defined as 24 consecutive months without menses before Screening, with a follicle stimulating hormone [FSH] level in the postmenopausal range according to the laboratory used at Screening); FSH to be performed at the discretion of the Investigator in consultation with the Medical Monitor.
7. Females of child-bearing potential (FCBP) must agree to practice a highly effective method of contraception throughout the study and for 5 months after the last dose of investigational product (IP). Acceptable methods of birth control in this study are the following:

   * Combined hormonal (containing oestrogen and progestogen) contraception, which may be oral, intravaginal, or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable or implantable
   * Placement of an intrauterine device or intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomised partner
   * Sexual abstinence
8. Male subjects must:

   1. Practice true abstinence (which must be reviewed on a monthly basis and source documented) or agree to use a latex condom during sexual contact with FCBP while participating in the study until 5 months after the last dose of IP.
   2. Agree to refrain from donating sperm during the study until 5 months after the last dose of IP.

   Periodic abstinence (calendar, symptothermal, postovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea method are not acceptable methods of contraception. Female condom and male condom should not be used together.
9. Subjects must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted, and must be able to comply with the requirements of the study, including the study visit schedule and other protocol requirements. Must be able to communicate with the Investigator and

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical history/condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever was longer).
5. Subject has a history of infection within 30 days of dosing on Day 1.
6. Subject has a history of drug or alcohol abuse (as defined by the investigator), or addiction within 6 months prior to Screening.
7. Subject has used any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, electronic cigarettes, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 3 months prior to Day 1 and during the study.
8. Subject has a positive urine drug test including cotinine, or positive alcohol urine or breath test at Screening or on Day -1.
9. Subject has donated greater than 400 mL of blood within 60 days prior to Day 1.
10. Subject has a positive serum test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV).
11. Subject has a history of clinically significant allergic reaction to any drug, biologic, food, or vaccine.
12. Subject has a history of major immunologic reaction (such as anaphylactic reaction, anaphylactoid reaction, or serum sickness) to any IgG-containing agent.
13. Subject fails or is unwilling to abstain from strenuous physical activities for at least 24 hours prior to dosing (Day 1) and throughout the study
14. Subject has tattoos (> 25% of their body) or other skin markings (eg, scars) that, in the opinion of the investigator, would prevent visualization of dermatologic changes due to study treatment
15. Subject has been diagnosed with or is being treated for a parasitic/helminthic infection or subject has systemic or diarrheal illness following travel or residence in endemic areas of parasitic/helminthic infections, history of clinical schistosomiasis, and history of travel to endemic areas within preceding 6 months.
16. Subject has a history of tuberculosis, listeriosis, or untreated parasitic infections.
17. Subject has a history of hereditary fructose intolerance.
18. Subject is, for any reason, deemed by the Investigator to be inappropriate for this study.
19. Subject has received any drug by injection within 30 days of Day 1.
20. Subject has poor peripheral venous access.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - AUC0-last | from pre-dose to up to Day 70
  Area under the concentration-time curve calculated from time zero to the last measured concentration
Pharmacokinetics - AUC0-∞ | from pre-dose to up to Day 70
  Area under the concentration-time curve calculated from time zero to infinity
Pharmacokinetics - Cmax | from pre-dose to up to Day 70
  Maximum observed concentration of drug
Pharmacokinetics - tmax | from pre-dose to up to Day 70
  Time to Cmax
Pharmacokinetics - t½ | from pre-dose to up to Day 70
  Terminal elimination half-life
Pharmacokinetics - CL/F | from pre-dose to up to Day 70
  Apparent clearance of drug from serum after extravascular administration
Pharmacokinetics - Vz/F | from pre-dose to up to Day 70
  Apparent volume of distribution during the terminal phase

SECONDARY OUTCOMES:
Adverse Events (AEs) | From the time the informed consent form (ICF) is signed and until 70 days after the last dose of CC-93538
  Number participants with adverse event
Immunogenicity profile for CC-93538 | from pre-dose to up to Day 70
  Positive or negative for the presence of antidrug antibodies against CC-93538 in blood

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tran, Pharm.D, Study Director — Celgene
Locations (1):
- Anaheim Clinical Trials, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/